CLINICAL TRIAL: NCT06252415
Title: Evaluation of Rapid First-line Genome Sequencing for Prenatal Diagnosis of Congenital Malformations in Comparison With Chromosomal Microarray and Exome Sequencing
Acronym: PRENATOMEultra
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: OLIVIER FAIVRE 2023
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Congenital Malformation
MeSH Terms: conditions — Congenital Abnormalities | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- parent-to-be: Pregnant women and the biological father
  Interventions: Biological: foetal amniotic fluid sample; Biological: blood samples; Other: semi-structured online interviews

INTERVENTIONS:
Biological: foetal amniotic fluid sample — At the inclusion visit, during the foetal samples taken for the CMA/ES as part of the care.
Biological: blood samples — 2 x 5ml blood EDTA tubes for both parents
Other: semi-structured online interviews — 25 included couples will be invited to take part in 2 semi-structured online interviews (by telephone or videoconference)

SUMMARY:
The management of congenital malformations (3% of pregnancies) by prenatal ultrasound represents a real medical challenge. Their prognosis is variable depending on the underlying aetiology. In France, prenatal diagnosis (PND) has long been based on imaging or infectious, metabolic, immunological or genetic investigations (karyotype, chromosomal microarray (CMA) and sequencing of targeted genes in some cases). About 70% of foetuses remain without an etiological diagnosis after these investigations. Exome (ES) and genome sequencing (GS) has revolutionized medical genetics, with a postnatal diagnostic rate of more than 40% for developmental disorders in the absence of clinical orientation and/or after a negative standard workup. In PND, trio-ES has been progressively introduced in several countries in a diagnostic approach to refine the prognosis and help couples to make decisions regarding the current pregnancy, but also for the subsequent family planning/counselling. However, the delay in the return of results, 3 to 4 weeks on average, is long for couples. Also, ES cannot detect some variants, like structural variants, accessible to GS, that may lead to additional diagnosis in 5 to 10% of cases.

Since 2013, the FHU TRANSLAD has been transferring ES in diagnosis for patients with rare diseases with developmental anomalies, by deploying different pilot projects. In PND, our team was the first in France to propose a national research project, AnDDI-Prenatome, supported by the AnDDI-Rares health network, to evaluate the feasibility of analyzing ES and delivering results in less than 4 weeks in the context of congenital malformations (PMID:37035737). The teams were able to demonstrate the feasibility of prenatal ES implementation, with on overall diagnostic yield of 41% (37/89) when ES was used as a first-line test and 31% (19/61) when used after a normal CMA. This experience has enabled the implementation of ES in routine diagnosis, with an offer for the French hospitals. Our team now coordinates the DPNI-Exome trial (interregional PHRC; NCT05182242), comparing non-invasive and invasive approaches for fetal ES in PND when foetal ultrasound signs are discovered.

Our team now wishes to evaluate the diagnostic yield and the percentage of results delivery in less than 7 days of rapid trio-GS in case of ultrasound signs, to reduce the delay of results, but also possibly increase the rate of PND. In addition, information concerning the efficiency of rapid trio-GS as well as technical hurdles associated with its implementation will permit the development of national guidelines.

This is a question of outmost importance from an international scientific point of view because currently only six publications have proposed the use of the rapid prenatal GS, while around seventy studies report an experience of prenatal ES. Five of these six publications were from China, sometimes retrospective, with no or limited information regarding the methods, inclusion criteria, delays, nor difficulties encountered, and often a low number of included patients. The efficiency cannot be deducted from these publications. The proposed study should answer if rapid trio-GS could be implemented in routine PND in France.

The team is committed to assessing the impact of new reproductive technologies on couples. It has already carried out longitudinal qualitative studies, in the DPNI-Exome study, which showed the difficulties couples face when waiting for different results, delivered in different timeframes. GS makes it possible to offer only one unique test, which could answer the parents' questions. The team do their best to ensure that the results are delivered very quickly, but the psychologists mentioned that waiting for the results gives the couple sufficient time to realise the discovery of ultrasound signs, and the possible impact on the pregnancy prognosis. It is therefore important to assess couples' perceptions and satisfaction with a single test, which is quicker than what is offered in the standard care, and to evaluate whether the time needed to obtain the results is sufficient for their decision-making. This could be assessed by semi-directive interviews.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancies (17 - 34 weeks of gestation (WG)) with US anomalies namely either i) two major anomalies, ii) one major and one minor anomalies, or iii) one anomaly (major or minor) with a strong suspicion of genetic cause (such as corpus callosum anomaly);
* Couples for whom an etiological diagnosis could modify the pregnancy outcome and/or the pre and/or postnatal management;
* Pregnant women who receive invasive prenatal sampling for ES+CMA;
* Sufficient quantity of amniotic fluid to collect an additional sample for GS;
* Possibility of blood samples from the pregnant woman and the biological father;
* Written consent for genetic analysis from pregnant woman and biological father of foetus;
* Provision of signed and dated of both parents' consent form for the study.

For the exploratory qualitative objective/endpoint:

- A least one member of the couple willing to accept 2 telephone or video consultations, and able to speak and understand French.

Exclusion Criteria:

* Refusal of the pregnant woman or biological father to participate in the study; or refusal to collect blood samples from one or both parents;
* Pregnancy before 17 WG or after 34 WG (to limit the risk of reporting results after birth);
* Isolated increase nuchal translucency on ultrasound;
* Couples for whom an etiological diagnosis would not modify the pregnancy outcome;
* Pregnant woman and biological father not affiliated to a social security system or not beneficiaries of such a system;
* Pregnant woman and/or biological father who are protected and unable to understand the protocol and express their consent;
* Pregnant women and/or biological fathers under legal protection (guardianship, tutorship) or to a court order

For the exploratory qualitative objective/endpoint:

- The two members of the couple unable to carry out two one-hour telephone interviews in French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women and the biological father, eligible for the study, will be identified by an investigator at a genetic consultation dedicated to the proposal of prenatal CMA/ES within one of the rare disease reference centers of the AnDDI-Rares health and CPDPN networks declared in the study.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
the delay between sampling and the delivery of the results of the rapid GS strategy in less than 7 days | Through study completion, on average of 9 month
  In order to assess the interest of rapid GS as a first-line tool, we will consider two main co-criteria
the identification of one or more class 4 or 5 variant(s) that explain the ultrasound manifestations, and validated during a specific MultiDisciplanary Meeting (MDM) | Through study completion, on average of 9 month
  In order to assess the interest of rapid GS as a first-line tool, we will consider two main co-criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France